CLINICAL TRIAL: NCT02802605
Title: Randomized and Controlled Trial on the Safety and Efficacy of Bemiparin in the Prevention of Thrombotic Events in Hospitalized Cirrhotic Patients
Brief Title: Safety and Efficacy of Bemiparin in the Prevention of Thrombotic Events in Hospitalized Cirrhotic Patients
Acronym: BEMI-2015
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BEMI-2015
Record Dates: First submitted 2016-05-31; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Cirrhosis and Coagulation
MeSH Terms: conditions — Fibrosis; Thrombosis | interventions — bemiparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bemiparin (Experimental): Bemiparin 3.500 U, once a day during hospitalization
  Interventions: Drug: Bemiparin
- No drug (No Intervention): Clinical practice as usual

INTERVENTIONS:
Drug: Bemiparin — Bemiparin subcutaneus administration
  Arms: Bemiparin

SUMMARY:
Prospectively evaluation of the incidence of thromboembolic events in hospitalized cirrhotic patients. 2. Efficacy and safety of use of bemiparin in preventing peripheral and portal thrombosis. 3. Monitoring antiXa levels.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: To evaluate the safety of prophylactic anticoagulation Bemiparina (HIBOR®) for the prevention of peripheral and portal vein thrombosis in cirrhotic patients with prolonged hospitalization.

Secondary objectives are the following:

1. To evaluate the incidence of thrombotic events in hospitalized cirrhotic patients.
2. To evaluate the efficacy of low molecular weight heparin (HIBOR 3.500UI) in preventing thrombotic events in hospitalized cirrhotic patients.
3. To identify risk factors for development of portal vein thrombosis and deep vein thrombosis in hospitalized patients.
4. Evaluate the morbidity and mortality associated with thromboembolic events.
5. Evaluate prophylactic anticoagulation levels by determining antiXa and antithrombin III.
6. To study the expression profile and functionality of Toll-like receptors as factors intimately involved in the inflammatory response, as well as the variability of different serum markers associated with proinflammatory state: I-FABP / IL6-IL8 / NO, endothelin and LPS-binding protein.
7. Evaluate the effect on liver fibrosis (by Fibroscan®) and serum TGF
8. Evolution of hepatocellular function estimated by the scores of Child-Pugh and MELD.

ELIGIBILITY:
Inclusion Criteria:

1. Liver cirrhosis of any etiology diagnosed by previous biopsy or clinical, laboratory and sonographic criteria
2. Hospital admission at least 3 days, because of decompensated liver disease (ascites, encephalopathy, controlled gastrointestinal bleeding, spontaneous bacterial peritonitis)
3. signed written consent
4. Women of child-bearing age use effective contraception

Exclusion Criteria:

1. Age <18 and >80 years
2. contraindication to treatment with heparins
3. uncontrolled hemorrhage
4. Any comorbidity involving a therapeutic limitation and / or a life expectancy <6 months
5. concomitant antiplatelet therapy (aspirin, clopidogrel, ticlopidine, dipyridamole, sulfinpyrazone, dextran 40, or other anticoagulants
6. and continued concomitant NSAIDs, salicylates, corticosteroids
7. existence of clinically significant esophageal varices / severe gastropathy of portal hypertension without their having been previously treated with primary / secondary prophylaxis (endoscopic variceal ligation / non cardioselective beta blockers)
8. Refusal to participate in the study, or to sing informed consent
9. Pregnancy or lactation
10. HIV infection
11. platelet count <20,000 platelets / dl
12. renal clearance below 30ml / min
13. portal vein thrombosis or peripheral thrombosis diagnosed at admission
14. presence of procoagulant factor previously known

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with bleeding and liver toxicity under Bemiparin treatment (HIBOR®) for the prevention of DVT / portal vein thrombosis. | 90 days
  The bleeding will be classificated in two grades ( mild/ severe) and hepatoxicty were asses according to NCI CTCAE Version 3.0

SECONDARY OUTCOMES:
Number of thrombotic events in cirrhotic hospitalized patients | 90 days

IPD SHARING:
Plan to Share IPD: No